CLINICAL TRIAL: NCT02946164
Title: Advancing HIV Prevention and Linkage to Care Among MSM With Gamification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: AIDS Healthcare Foundation (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH106359 (NIH)
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comparison: Standard of Care (No Intervention): Standard services available to all men at AHF Wellness Centers.
- Intervention: 'Stick To It' Intervention (Active Comparator): Behavioral intervention.
  Interventions: Behavioral: Stick To It

INTERVENTIONS:
Behavioral: Stick To It — The intervention is a prize system linked to points earned through online and real-world activities designed to incentivize young MSM to test for HIV and STIs every three months. Participants receive points for pre-determined activities, such as: answering online quizzes, inviting friends to participate, and getting tested for HIV/STIs. Points are redeemable in person at two AIDS Healthcare Foundation Men's Wellness Centers, where participants will be able to exchange their points for gumballs from a gumball machine; different color combinations of gumballs correspond to prizes of different values. Participants are reminded to get tested regularly via SMS messages; in addition, they can check when their next test is due by checking their testing timer on the stick2it.org website.
  Arms: Intervention: 'Stick To It' Intervention

SUMMARY:
This study is a pilot evaluation of 'Stick To It', a behavioral intervention based on the concept of gamification. The objective of the program is to encourage young men who have sex with men (MSM) to be regularly screened for HIV and sexually transmitted infections (STIs) and to adopt safer sexual behaviors, with the ultimate goal to decrease HIV and STI incidence. Gamification is the application of game elements, like points, badges, and rewards, to non-game settings.

DETAILED DESCRIPTION:
The investigators will conduct a quasi-experimental pilot study of 'Stick To It', a prevention intervention that uses gamification principles and mechanics. The intervention includes an online timer that reminds men to get tested, online quizzes, and peer recruitment; these activities are awarded with points redeemable for chances at prizes at participating clinics. The intervention was designed based on findings from interviews with health staff and focus groups with young MSM, and with input from a gamification consultant. The primary hypothesis is that the intervention will increase repeat HIV/STI testing among young MSM. The intervention will be implemented at two STI clinics in Oakland and Los Angeles, California in 2-week intervals for six months. The investigators will review medical records of exposed and unexposed young MSM attending the same STI clinics to compare uptake of quarterly HIV testing and self-reported behavior after six months.

ELIGIBILITY:
Inclusion Criteria:

* 18-26 years of age
* male
* self-identify as gay / bisexual / queer
* willing and able to provide informed consent to join the Stick To It program
* resident in one of several zip code areas surrounding the clinic

Exclusion Criteria:

* Not a resident of one of included zip code areas

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2016-10; Primary Completion 2017-10-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Repeat HIV Testing | 6 months
  The number of men in the intervention who receive ≥1 additional HIV tests over 6 months of follow-up

SECONDARY OUTCOMES:
HIV-related risk behavior | 6 months
  We will determine the number of reported sex partners, the prevalence and frequency of unprotected anal intercourse with a partner of opposite or unknown status in the past 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandra I McCoy, PhD, Principal Investigator — Assistant Adjunct Professor
Locations (2):
- United States (2):
  - AHF Hollywood Wellness Center, Los Angeles, California
  - AHF Wellness Center Oakland, Oakland, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mejia CM, Acland D, Buzdugan R, Grimball R, Natoli L, McGrath MR, Klausner JD, McCoy SI. An Intervention Using Gamification to Increase Human Immunodeficiency Virus and Sexually Transmitted Infection Screening Among Young Men Who Have Sex With Men in California: Rationale and Design of Stick To It. JMIR Res Protoc. 2017 Jul 17;6(7):e140. doi: 10.2196/resprot.8064. PMID 28716771